CLINICAL TRIAL: NCT05141526
Title: Non-restrictive Approach to Facilitate Appetite Control and Long-term Body Weight Loss in Individuals With Obesity: Can we do Better?
Brief Title: Satiating Diet, Appetite Control and Body Weight Loss in Individuals With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Vicky Drapeau, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAT-2-129796
Record Dates: First submitted 2021-09-20; First posted 2021-12-02 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Weight Loss; Weight Maintenance; Appetite Control
MeSH Terms: conditions — Weight Loss | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: (1) non-restrictive, satiating intervention (P1) followed by a continuation of this intervention (P2); (2) conventional restrictive intervention (-500 kcal/d) (P1) followed by a non-restrictive satiating intervention (P2); (3) control group that follows minimal healthy guidelines (P1) followed by recommended weight maintenance strategies (P2). *P1=phase 1; P2=phase 2
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding participants is not possible due to the nature of the interventions. Individuals independent from the study and blinded to groups (e.g. statistician), will conduct the randomization and analyses while a research assistant, instructed not to discuss treatments with participants, will conduct the testing sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-restrictive satiating intervention (Experimental): The non-restrictive satiating intervention will include guidelines and recipes to prepare highly satiating meals that will be low in energy density and glycemic index and high in protein, polyunsaturated fats, vitamins and minerals (e.g. calcium), and certain constituents of spices (e.g. capsaicin).
  Interventions: Other: Non-restrictive satiating intervention
- Conventional restrictive intervention + non-restrictive satiating intervention (Experimental): Conventional restrictive intervention consisting of a -500 kcal/d calorie deficit (P1) followed by a non-restrictive satiating intervention (P2)
  Interventions: Other: Conventional restrictive intervention + non-restrictive satiating intervention
- Minimal healthy guidelines (Placebo Comparator): Considering recommendations from the latest Canadian Obesity Guidelines, the control group will receive a minimal intervention based on the Canada's Food Guide for Healthy Eating
  Interventions: Other: Control group

INTERVENTIONS:
Other: Non-restrictive satiating intervention — Diet group containing satiating foods
  Arms: Non-restrictive satiating intervention
Other: Conventional restrictive intervention + non-restrictive satiating intervention — Diet group with a calorie deficit during the first phase followed by a diet containing satiating foods in the second phase
  Arms: Conventional restrictive intervention + non-restrictive satiating intervention
Other: Control group — This group will receive minimal healthy guidelines
  Arms: Minimal healthy guidelines

SUMMARY:
The objective of this study is to evaluate (1) the effect of a non-restrictive satiating intervention on appetite control, body weight loss and maintenance; and (2) determine whether switching to a non-restrictive satiating intervention following a conventional restrictive intervention can prevent increases in appetite and attenuate body weight regain usually observed after weight loss in men and women living with obesity. This is an 18-month, randomized, controlled, parallel weight loss [Phase 1 (P1): 6 months] and maintenance trial [Phase 2 (P2): 12 months] with three groups (n=234 men and women): (1) non-restrictive, satiating intervention (P1) followed by a continuation of this intervention (P2); (2) conventional restrictive intervention (-500 kcal/d) (P1) followed by a non-restrictive satiating intervention (P2); (3) control group that follows minimal healthy guidelines (P1) followed by recommended weight maintenance strategies (P2). All groups will be controlled for physical activity and sleep patterns. The non-restrictive satiating intervention will include guidelines and recipes to prepare highly satiating meals that will be low in energy density and glycemic index and high in protein, polyunsaturated fats, vitamins and minerals (e.g. calcium), and certain constituents of spices (e.g. capsaicin). Measurements at baseline (week 0), after P1 and P2 will include the following primary outcomes: appetite control, weight loss and maintenance; and secondary outcomes: body composition, physiological, psycho and neurobehavioural and health-related variables. Follow-ups will be done by a dietitian every 2 weeks during P1 and once a month during P2.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a BMI ≥30 and <40 kg/m2
* aged between 18-50 years
* waist circumference >102 cm in men and >88 cm in women.

Exclusion Criteria:

* taking medications that could influence appetite or body weight (e.g. thyroid replacement therapy, sulfonylureas and glucocorticoids)
* being treated with insulin for type 2 diabetes
* large body weight fluctuations (>4 kg over last two months)
* characterized by high restraint behaviour (score >12, measured with the TFEQ)
* history of an eating disorder (e.g. binge eating disorder) using the EDE questionnaire
* performing >150 min of moderate-vigorous intensity physical activity/week
* use of nutritional supplements (multivitamins, calcium, protein, fibre); 8) smoking, drugs or alcohol (>2 drinks/d)
* consumption of >5 cups of coffee/d
* (pre)menopausal or pregnant women
* diagnosis of chronic diseases, acute infections or gastric problems (e.g. ulcers)
* food allergies/intolerances to ingredients/foods in the satiating intervention
* having a pacemaker (for fMRI)
* taking sedatives or sleeping pills
* symptoms of depression (>20 on the BDI).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The research questions will take into account sex and gender as we consider: (i) restrictive and non-restrictive approaches that may have different impacts on body weight between men and women; and (ii) the impact of these interventions may have different outcomes on behavioural and psychosocial variables. Therefore, participants may be able to indicate their gender identity.
Enrollment: 234 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | 6 months
  Body weight loss (kg) after Phases 1 and 2
Body composition | 6 months
  Body fat (using dual x-ray absorptiometry)
Hunger/Satiety | 6 months
  using a visual analogue scale and measured in mm
Energy intake | 6 months
  measured at an ad libitum meal in kilocalories

SECONDARY OUTCOMES:
Stress | 18 months
  State-Trait Anxiety Inventory
Anxiety | 18 months
  Perceived Stress Scales
Eating Behaviours | 18 months
  Three Factor Eating Behaviour Questionnaire
Depression Symptoms | 18 months
  Beck Depression Inventory
Lipids (HDL-cholesterol, LDL-cholesterol, triglycerides, total cholesterol) | 18 months
  measured in mmol/L
Blood pressure | 18 months
  mmHg
Diet satisfaction | 18 months
  Diet Satisfaction Questionnaire (scale: strongly disagree to strongly agree)
neurobehavioural variables | 6 months
  brain anatomy and activity in response to food cues (using fMRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education, Québec, Quebec, Canada